CLINICAL TRIAL: NCT04485273
Title: Effect of Dexmedetomedine in Subtenon's Block on Emergence Agitation in Pediatric Strabismus Surgery Under Sevoflurane Anesthesia
Brief Title: Effect of Dexmedetomedine in Subtenon's Block on Emergence Agitation in Pediatric Strabismus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sameh Fathy (Other)
Responsible Party: Sponsor-Investigator, Sameh Fathy, Lecturer of anesthesia, ICU & pain management; Faculty of Medicine, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dexmedetomedine and agitation
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Emergence Agitation
Keywords: Dexmedetomedine; Subtenon's Block
MeSH Terms: conditions — Emergence Delirium | interventions — Laryngeal Masks; Sevoflurane; Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomedine Group (Active Comparator): Laryngeal mask airway is inserted and anesthesia is maintained with sevoflurane. Subtenon's block is performed and local anesthetic solution is injected, in addition to dexmedetomedine.
  Interventions: Device: Laryngeal Mask Airway; Drug: Sevoflurane; Procedure: Subtenon's Block; Drug: Local Anesthetic Solution and Dexmedetomedine
- Control Group (Placebo Comparator): Laryngeal mask airway is inserted and anesthesia is maintained with sevoflurane. Subtenon's block is performed and local anesthetic solution is injected.
  Interventions: Device: Laryngeal Mask Airway; Drug: Sevoflurane; Procedure: Subtenon's Block; Drug: Local Anesthetic Solution

INTERVENTIONS:
Device: Laryngeal Mask Airway — Capnography connected to laryngeal mask airway is introduced after adequate jaw relaxation and oral airway tolerance; its size is chosen according to the body weight of the child.
  Other Names: Supraglottic Airway Device
Drug: Sevoflurane — Sevoflurane in air/oxygen mixture of 40% is titrated to achieve adequate depth of anesthesia.
  Other Names: Inhalational Anesthesia
Procedure: Subtenon's Block — Subtenon's block is performed in the eye undergoing surgery under sterile conditions where a 19-gauge curved blunt metallic cannula (25 mm) is inserted into sub-tenon's space.
  Other Names: Regional Eye Block
Drug: Local Anesthetic Solution and Dexmedetomedine — The local anesthetic solution is injected with a dose of 0.5% bupivacaine (0.08 ml/kg), in addition to dexmedetomedine (0.5 μg /kg)
  Other Names: Marcaine and Precedex
  Arms: Dexmedetomedine Group
Drug: Local Anesthetic Solution — The local anesthetic solution is injected with a dose of 0.5% bupivacaine (0.08 ml/kg).
  Other Names: Marcaine
  Arms: Control Group

SUMMARY:
The study is conducted to evaluate the effects of dexmedetomedine in subtenon's block in conjunction to general anesthesia under sevoflurane anesthesia on emergence agitation, intraoperative hemodynamic stability, postoperative pain, nausea and vomiting in patients undergoing strabismus surgery.

DETAILED DESCRIPTION:
Emergency agitation is a clinical status of postoperative excitement or emergence delirium when the patient is awake but is disorientated. It is described as mental disturbances that consist of confusion, hallucinations and delusions which is manifested by restless involuntary physical activity and thrashing about the bed. Its incidence has been observed especially in pediatric ophthalmology care units due to many factors such as pain, mental status, time of operation, age, lack of ability to see outside, and a history of previous hyperthermia. Strabismus surgery is one of the most frequently performed pediatric ocular operations. However, it can cause unfavorable side effects during intraoperative and postoperative periods. Typically, the major problems associated with strabismus surgeries include increased risk of the oculocardiac reflex, postoperative pain, nausea and vomiting. Subtenon's block is one of the regional anesthetic techniques used in ocular surgery. Dexmedetomidine has been used as an adjuvant to local anesthetics for regional anesthesia in various clinical fields including the subtenon's block.There is evidence that dexmedetomidine decreases the incidence of agitation after sevoflurane anesthesia in children undergoing different surgical procedures. Therefore, this study is conducted to evaluate the effect of dexmedetomedine in subtenon's block on emergence agitation in pediatric strabismus surgery under sevoflurane anesthesia.

This prospective, randomized, clinical study includes 100 children who are scheduled for elective strabismus surgery under general surgery in Mansoura ophthalmology center. Informed written consent is obtained from parents of all subjects in the study after ensuring confidentiality.The study protocol is explained to parents of all patients in the study who are kept fasting prior to surgery. Patients are randomly assigned to two equal groups according to computer-generated table of random numbers using the permuted block randomization method.The collected data are coded, processed, and analyzed using SPSS program. All data are considered statistically significant if P value is ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) I and II patients.
* Scheduled for strabismus surgery.

Exclusion Criteria:

* Parental refusal of consent.
* Contraindication to use of supraglottic airway device as gastroesophageal reflux and oropharyngeal pathology.
* Hyperactive airway disease or respiratory diseases.
* Children with developmental delays, mental or neurological disorders.
* Bleeding or coagulation diathesis.
* History of known sensitivity to the used anesthetics.
* Previous surgery in the same eye

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in postoperative emergence agitation scale | Up to 30 minutes after surgery
  Agitation is assessed using the 5- step Cravero scale (1-5) every five minutes from awakening and for 30 minutes.(1:Obtunded with no response to stimulation, 2:Asleep but responsive to movement or stimulation, 3:Awake and responsive, 4:Crying, 5:Thrashing behaviour that requires restraint)
Emergence time | Up to 30 minutes after surgery
  Emergence time (min) is recorded; from the discontinuation of sevoflurane to the first response on verbal command.

SECONDARY OUTCOMES:
Changes in heart rate | Up to the end of the surgery
  Heart rate (beat/min) is recorded at five-minute intervals until the end of the surgery.
Changes in mean arterial blood pressure | Up to the end of the surgery
  Blood pressure (mmHg) is recorded at five-minute intervals until the end of the surgery.
Incidence of oculocardiac reflex | Up to the end of the surgery
  If there is dysrhythmia or rapid reduction in HR by more than 25% from the baseline, it is considered as an oculocardiac reflex.
Changes in pain scores | Up to 24 hours after the procedure
  Pain score from 0 to 10 (0 = no pain and 10 = the worst imaginable pain) is assessed every two hours up to 24 hours after the procedure.
Total analgesic requirements of paracetamol | Up to 24 hours after the procedure
  The amount of paracetamol consumption given as a rescue analgesia to patients is measured all over the 24 hours.
First analgesic request | Up to 24 hours after the procedure
  The time of the first analgesic request for paracetamol is recorded.
Incidence of postoperative nausea and vomiting | Up to 24 hours after the procedure
  Incidence of postoperative nausea and vomiting is assessed up to 24 hours after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh M El-Sherbiny, MD, Principal Investigator — Mansoura Faculty of Medicine
Locations (1):
- Department of Anesthesia, Mansoura University Hospitals, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No